CLINICAL TRIAL: NCT03610932
Title: Vitamin C Supplementation to Improve EIB in College Student-Athletes
Brief Title: Vitamin C & Exercise Induced Bronchoconstriction (EIB)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY00140641
Record Dates: First submitted 2018-06-07; First posted 2018-08-01 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Exercise-induced Bronchospasm
MeSH Terms: conditions — Asthma, Exercise-Induced | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental): Participants will ingest 3 (500 mg) capsules of Vitamin C each day for 2 weeks.
  Interventions: Dietary Supplement: Vitamin C
- Placebo (Active Comparator): Participants will ingest a matched capsule for size and color to the Vitamin C supplement.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — Taken as 3 500mg capsules.
  Arms: Vitamin C
Other: Placebo — Taken as 3 500mg capsules.
  Arms: Placebo

SUMMARY:
The purpose of this research is to assess the association between diet and pulmonary function during standardized EIB testing. Determine the effect of Vitamin C supplementation on airway inflammatory markers and bronchoconstriction after a standardized EIB test compared to usual diet and placebo control.

DETAILED DESCRIPTION:
This study will use a double-blind, randomized, cross-over design with subjects serving as their own controls. This study will be conducted over a consecutive five-week period.

All subjects will be asked to discontinue taking their short- and long-acting beta-agonist medication 12 and 24 hours respectively prior to data collection. Also, all subjects will be asked to refrain from caffeine, physical activity, and NSAID use 24 hours prior to testing. In addition all subjects will be asked to abstain from taking any vitamin supplement during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Student or student-athlete who has tested positive for EIB
* Able to communicate in English

Exclusion Criteria:

* Forced expiratory volume in 1 second (FEV1) < 70% of predicted, cardiac history,
* Current respiratory infection
* > 10 pack year history of smoking
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
Change in airway inflammatory biomarkers | Change from Baseline to End of Week 5
  Urinary concentrations of cysteine leukotrienes (LTC4-LTE4), prostaglandin (9α,11β-PGF2), and creatinine will be measured.

SECONDARY OUTCOMES:
Change in quality of life: asthma quality of life questionnaire (AQLQ) | Change from Baseline to End of Week 5
  Asthma specific quality of life will be measured by the validated asthma quality of life questionnaire (AQLQ). The AQLQ includes 32 separate responses within 4 domains: activity limitation (11 items), symptoms (12 items), emotional function (5 items), and environmental stimuli (4 items). Each response option is based on a 7-point scale, where 1 represents maximal impairment and 7 indicates no impairment. Scores for the four domains and overall score are computed as averages of the item scores. The minimal important difference for overall and each domain, has been determined to be a change in score of 0.5 per item.
Dietary Intake Questionnaire | Change from Baseline to End of Week 5
  Baseline dietary intake will be assessed by the National Cancer Institute's Diet Health Questionnaire II (DHQ II). It consists of 134 food items and 8 dietary supplement questions. It calculates the Healthy Eating Index (HEI) that is a measure of diet quality. Scores range from 0 to 100. The higher the score the healthier the diet.
Cardiorespiratory Fitness | Baseline
  Cardiorespiratory fitness will be assessed during the EIB test by an integrated metabolic measurement system that will be used for measurement of oxygen consumption. The metabolic cart will be set to produce a 15-second average of the data collected during gas analyses for all tests.
Pulmonary function testing | Change from Baseline to End of Week 5
  The outcome will measure the change in the first second of forced expiration (FEV1).

CONTACTS AND LOCATIONS:
Overall Officials: Dave Burnett, PhD, RRT, AE-C, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States